CLINICAL TRIAL: NCT05128695
Title: Long-term Public Health Consequences of Covid-19-- Physical, Mental and Social Health
Brief Title: Public Health Consequences of Covid-19
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Public Health Service South Limburg (Other Government)
Collaborators: Maastricht University (Other); Center for Integrated Rehabilitation and Organ Failure Horn (Other); National Institute for Public Health and the Environment (RIVM) (Other Government); Public Health Service North Limburg, Netherlands (Other Government)
Responsible Party: Principal Investigator, Nicole Dukers-Muijrers, Senior epidemiologist, associate professor, Public Health Service South Limburg
Other Study IDs: 2021-2884
Record Dates: First submitted 2021-11-17; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
Keywords: Covid-19; Longcovid; Mental health; Loneliness; Depression; Fatigue; Social health; Care consumption; Public Health
MeSH Terms: conditions — COVID-19; Psychological Well-Being; Depression; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid-19 positive: Adults who tested Covid-19 positive
  Interventions: Other: there is no intervention; the study is observational
- Covid-19 negative: Adults who tested Covid-19 negative
  Interventions: Other: there is no intervention; the study is observational

INTERVENTIONS:
Other: there is no intervention; the study is observational — there is no intervention; the study is observational

SUMMARY:
Aim of this observational study is to improve our understanding of the impact of Covid-19 on health. By an online questionnaire at least 60.000 people are invited by email to participate. Invited are those people who tested for Covid-19 at the Public Health Service South Limburg since June 2020. Participants are followed over time (open cohort), to study impact on health, that is physical health, mental health, and social health (longcovid and other conseauences). Also, the socioeconomic impact is studied, as on work and education. And the consequences for health-care consumption; it also includes aspects as coping, stigma and lifestyle. All focused to understand the impact of Covid-19, in relation to health, and to gain information for promoting positive health and improving prevention and care.

DETAILED DESCRIPTION:
Design: Prospective observational cohort study Mode of study: Online questionnaires Timing: Baseline starting nov. 2021; with regular follow-up measurements Measures: A great range of health-associated factors, all self-reported including a range of physical, mental and social health aspects.

A range of structural and functional social netwok aspects Various measures on Covid-19 testing and vaccination Various measures on lifestyle behavior. And other measures that are interlinked with health-factors (such as coping, stress, and sociostructural factors) Analyses: Quantitative data are collected prospectively, and assessed using the appropriate data-analyses methods. Thee include for example epidemiological statistical methods, and social network methodology.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Having recieved an online invitation to participate by an email with the study information and questionnaire link, which is send based on the email that was provided to the Public Health service upon testing for Covid-19 at the public health service south Limburg

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults (aged 18+) who received a test for Covid-19 from the public health service south limburg from june 2020 onward, and who provided an email adress can be selected to be invited in this study.
  This includes all people who tested positive. This includes a representative fraction (based on month of testing, age-group, sex, and region of residence) of those who tested negative.
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Longcovid | Change from the baseline questionaire up to 4 years thereafter, assessed at regular intervals (3,6,12 monthly) (note that at baseline, also historical information is collected from the participants)
  The symptoms that are defined by the WHO-definition of longcovid plus exploratory (data-driven--can include symptoms not in the current WHO-definition)
Mental health | Change from the baseline questionaire up to 4 years thereafter, assessed at regular intervals (3,6,12 monthly) (note that at baseline, also historical information is collected from the participants)
  Negative health-outcomes related to mental health such as depression (assessed by PRQ9 scale)
Social health | Change from the baseline questionaire up to 4 years thereafter, assessed at regular intervals (3,6,12 monthly) (note that at baseline, also historical information is collected from the participants)
  Negative health outcomes related to social health, such as loneliness (assessed by de Jong-Gierveld scale)
Physical health | Change from the baseline questionaire up to 4 years thereafter, assessed at regular intervals (3,6,12 monthly) (note that at baseline, also historical information is collected from the participants)
  Negative health-outcomes related to physical health such as chronic non communicable disease (assessed upon self-report on a checklist of conditions present)
Positive health and resilience | Change from the baseline questionaire up to 4 years thereafter, assessed at regular intervals (3,6,12 monthly)
  Experienced general health (5-point scale ECHI)

SECONDARY OUTCOMES:
Productivity | Change from the baseline questionaire up to 4 years thereafter, assessed at regular intervals (3,6,12 monthly)
  Socioeconomic impact on work and education (various scales)
Adversity | change from the baseline questionaire up to 4 years thereafter, assessed at regular intervals (3,6,12 monthly)
  Stigma and coping strategies related to Covid-19 adverse consequences

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Dukers-Muijrers, PhD, Study Chair — Public Health Service South Limburg
Locations (1):
- Public Health Service South Limburg, Geleen, South Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Coded data from this study will be made available for other researchers in due time

REFERENCES:
- [Derived] Pagen DME, van Bilsen CJA, Brinkhues S, Van Herck M, Konings K, den Heijer CDJ, Ter Waarbeek HLG, Spruit MA, Hoebe CJPA, Dukers-Muijrers NHTM. Prevalence of Long-term Symptoms Varies When Using Different Post-COVID-19 Definitions in Positively and Negatively Tested Adults: The PRIME Post-COVID Study. Open Forum Infect Dis. 2023 Sep 18;10(10):ofad471. doi: 10.1093/ofid/ofad471. eCollection 2023 Oct. PMID 37885796
- [Derived] Pagen DME, van Bilsen CJA, Brinkhues S, Moonen CPB, Van Herck M, Konings K, den Heijer CDJ, Mujakovic S, Ter Waarbeek HLG, Bouwmeester-Vincken N, Vaes AW, Spruit MA, Hoebe CJPA, Dukers-Muijrers NHTM. Design and recruitment of a large-scale cohort study on prevalence, risk factors and impact evaluation of post-COVID-19 condition and its wider long-term social, mental, and physical health impact: The PRIME post-COVID study. Front Public Health. 2022 Dec 15;10:1032955. doi: 10.3389/fpubh.2022.1032955. eCollection 2022. PMID 36589958